CLINICAL TRIAL: NCT03139669
Title: Cultural Acceptability and Feasibility of HPV Cervical Self Collection Aided by Lay Navigators
Acronym: HPVhometest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Emma McKim Mitchell, PhD, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18473
Record Dates: First submitted 2016-01-27; First posted 2017-05-04 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Human Papilloma Virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPV home testing kit (Experimental): The procedures will be recruitment of under-screened women in Health Districts 1, 2 and 3 of Southwest Virginia to complete HPV home testing using self-collection kits distributed by lay navigators. Regardless of HPV positivity, all women will be provided with information about cervical cancer screening (locations, cost, etc.), and will be encouraged to complete Pap screening by a clinician.
  Interventions: Device: Viba collection brush

INTERVENTIONS:
Device: Viba collection brush — HPV home collection kit using the viba collection brush to collect cervical cells for HPV DNA testing.

SUMMARY:
Invasive cervical cancer incidence and mortality can be dramatically reduced through early detection and treatment, but many women do not complete screening at recommended intervals. Many low-income women in Virginia remain uninsured and are at significant risk of being medically underserved and failing to complete regular cervical cancer screening. At-home self-collection of specimens for HPV testing is an innovative approach that may increase access to cervical cancer screening in populations that do not participate in traditional clinic-based screening. The proposed community based participatory study aims to determine whether offering at-home self-collection for HPV testing through a lay navigator network is an acceptable and feasible method to increase access to cervical cancer screening for under-screened women in the Tobacco Footprint in rural far Southwest Virginia (Health Districts 1, 2 and 3). The procedures will be recruitment of under-screened women in Health Districts 1, 2 and 3 of Southwest Virginia to complete HPV testing using self-collection kits distributed by lay navigators. Regardless of HPV positivity, all women will be provided with information about cervical cancer screening (locations, cost, etc.), and will be encouraged to complete Pap screening by a clinician.

DETAILED DESCRIPTION:
The catchment area for the University of Virginia Health System and Emily Couric Clinical Cancer Center (EC4) extends throughout Southwest Virginia and into neighboring West Virginia, encompassing a portion of Appalachia. State-wide incidence of cervical cancer was 6.6 cases per 100,000 from 2005-2009, but variation exists county by county: Cumberland (Health District 2), Roanoke, and Southside were among those with the highest incidence. The significant decrease in cervical cancer incidence and mortality rates in the US and in Virginia since 1950 is directly attributed to increased early detection and screening. The Virginia Department of Health's Comprehensive Cancer Control Program found that patient level barriers to screening for women in this region include lower education, lower income, and lack of health insurance. Systems-level barriers in this region include decreased access to screening services, financial barriers, and transportation barriers. This study will assess a novel approach to addressing patient level and systems-level barriers to accessing cervical cancer screening in Virginia Health Districts 1, 2 and 3, and utilizes an innovative technology (self-collection for HPV testing) and delivery model (distributed by lay navigators).

Self-collection for HPV testing paired with a community health worker program is a model that has been found to have great utility in accessing at risk women in several rural and remote areas around the world. Community health workers often have training in a variety of health issues and conditions. Patient navigators trained in cervical cancer screening and treatment specifically have been utilized to understand patient barriers to in-clinic screening. The lay navigator program the investigators will work with in Virginia Health Districts 1, 2 and 3 involves cancer-specific training (including but not limited to cervical cancer training), and training on facilitating access to screening and treatment resources available in Health Districts 1, 2 and 3, as well as at the University of Virginia Health System. Lay navigators are therefore uniquely poised to provide education to women around the use of HPV self-collection, and to navigate women to in-clinic Pap screening, treatment, and support services as needed.

Reach of Current Lay Navigators Trained using the "Understanding Cancer" curriculum (developed by partners listed above), lay navigators in Russell County (Cumberland Health District) reported 312 encounters between 2/10/14 and 12/17/14 classified as "preventative" specific to breast cancer. Between 1/23/14 and 9/24/14, navigators across Lenowisco Health District provided 233 cancer-related encounters, including navigation services for 4 women diagnosed with cervical cancer. The lay navigator program has the potential to be a rich resources for community based research in Southwest Virginia.

Protocol Development Dr. Mitchell was a Co-I on the NCI-funded project P30CA044579 (PI: Thomas Loughran, MD, 2014-2015). Through this work, the investigators developed a list of key stakeholders, which will be consulted in Phases I and II of this study. Additionally, the community advisory board (CAB) of the Cancer Center Without Walls initiative will be consulted throughout protocol development.

Dr. Mitchell developed a collaboration with Dr. Jennifer S. Smith, Associate Professor of Epidemiology at the University of North Carolina at Chapel Hill. Dr. Smith and her research team have extensive experience and expertise with HPV screening and prevention, specifically exploring delivery models for HPV self-collection in medically underserved areas of North Carolina. Dr. Smith and the research team have conducted multiple previous studies assessing the acceptability, feasibility, and validity of HPV self-collection. Through these studies, the investigators have identified brush designs that are minimally invasive, well-accepted, and effective for self-collection and sample preservation media that is non-toxic, safe for mailing, and stable at a range of temperatures; and have developed well-validated, field-tested illustrated instructions for self-collection that are comprehensible to low-literacy women.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years old
* Female
* Live in southwest VA
* Not pregnant-self reported

Exclusion Criteria:

* History of Papanicolaou test in the last 3 years
* History of hysterectomy or pelvic radiation
* Co-testing (pap test and HPV test at the same time) in the last 5 years
* English speaking

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Mitchell, PhD, Principal Investigator — Faculty

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackerson K, Gretebeck K. Factors influencing cancer screening practices of underserved women. J Am Acad Nurse Pract. 2007 Nov;19(11):591-601. doi: 10.1111/j.1745-7599.2007.00268.x. PMID 17970859
- [Background] Arbyn M, Sasieni P, Meijer CJ, Clavel C, Koliopoulos G, Dillner J. Chapter 9: Clinical applications of HPV testing: a summary of meta-analyses. Vaccine. 2006 Aug 31;24 Suppl 3:S3/78-89. doi: 10.1016/j.vaccine.2006.05.117. PMID 16950021
- [Background] Arbyn M, Verdoodt F, Snijders PJ, Verhoef VM, Suonio E, Dillner L, Minozzi S, Bellisario C, Banzi R, Zhao FH, Hillemanns P, Anttila A. Accuracy of human papillomavirus testing on self-collected versus clinician-collected samples: a meta-analysis. Lancet Oncol. 2014 Feb;15(2):172-83. doi: 10.1016/S1470-2045(13)70570-9. Epub 2014 Jan 14. PMID 24433684
- [Background] Racey CS, Withrow DR, Gesink D. Self-collected HPV testing improves participation in cervical cancer screening: a systematic review and meta-analysis. Can J Public Health. 2013 Feb 11;104(2):e159-66. doi: 10.1007/BF03405681. PMID 23618210
- [Background] Gravitt PE, Belinson JL, Salmeron J, Shah KV. Looking ahead: a case for human papillomavirus testing of self-sampled vaginal specimens as a cervical cancer screening strategy. Int J Cancer. 2011 Aug 1;129(3):517-27. doi: 10.1002/ijc.25974. PMID 21384341
- [Background] Balasubramanian A, Kulasingam SL, Baer A, Hughes JP, Myers ER, Mao C, Kiviat NB, Koutsky LA. Accuracy and cost-effectiveness of cervical cancer screening by high-risk human papillomavirus DNA testing of self-collected vaginal samples. J Low Genit Tract Dis. 2010 Jul;14(3):185-95. doi: 10.1097/LGT.0b013e3181cd6d36. PMID 20592553
- [Background] Kobetz E, Kish JK, Campos NG, Koru-Sengul T, Bishop I, Lipshultz H, Barton B, Barbee L. Burden of Human Papillomavirus among Haitian Immigrants in Miami, Florida: Community-Based Participatory Research in Action. J Oncol. 2012;2012:728397. doi: 10.1155/2012/728397. Epub 2012 Mar 15. PMID 22619675
- [Background] Mandigo M, Frett B, Laurent JR, Bishop I, Raymondville M, Marsh S, Kobetz E. Pairing community health workers with HPV self-sampling for cervical cancer prevention in rural Haiti. Int J Gynaecol Obstet. 2015 Mar;128(3):206-10. doi: 10.1016/j.ijgo.2014.09.016. Epub 2014 Nov 11. PMID 25468050
- [Background] Ely GE, White C, Jones K, Feltner F, Gomez M, Shelton B, Slone S, Van Meter E, Desimone C, Schoenberg N, Dignan M. Cervical cancer screening: exploring Appalachian patients' barriers to follow-up care. Soc Work Health Care. 2014;53(2):83-95. doi: 10.1080/00981389.2013.827149. PMID 24483330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPV Home Testing Kit
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HPV Home Testing Kit
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 44.8 [31 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Smoking Status (Current Smoker) [Count of Participants; unit: Participants]
  Current Smoker | 28
  Non-Smoker | 17
Seen healthcare provider in last year (yes/no) [Count of Participants; unit: Participants]
  Have seen a healthcare provider in the last year | 30
  Have not seen a healthcare provider in the last year | 11
  Missing | 4

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of At-home Self-collection for HPV Testing Among Under-screened Women in Southwest Virginia.
Description: ACCEPTABILITY was measured through: uptake of self-collection kit (yes/n).
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Home Testing Kit
Number analyzed (Participants) | 45
Participants | 45

2. Secondary Outcome: Feasibility of Utilizing Lay Navigators to Offer At-home HPV Self-collection as a Strategy to Increase Cervical Cancer Screening Among Under-screened Women in Southwest Virginia.
Description: FEASIBILITY was measured by: uptake of self-collection kits (y/n), and whether that sample was sufficient for processing a result. If acceptability (uptake) was high but sufficiency of sample collection was low, there would be decreased feasibility of this approach.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Home Testing Kit
Number analyzed (Participants) | 45
Participants
  HPV self-collection kit uptake, sufficient sample to process a result | 42
  HPV self-collection kit uptake, insufficient sample collected to process a result | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HPV Home Testing Kit
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT03139669/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03139669/ICF_001.pdf